CLINICAL TRIAL: NCT01846754
Title: Prevalence of Fatigue and Its Related Factors in Hemodialysis Patients
Brief Title: Prevalence of Fatigue in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201302037RINC
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Hemodialysis Patients
Keywords: Hemodialysis; Fatigue; Muscle strength; Metabolomics
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human blood: 5c.c.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemodialysis patients

SUMMARY:
The prevalence of end stage renal disease in Taiwan was listed first all over the world. Fatigue, which makes patients unable to be competitive to play their functional roles, is one of the most bothersome symptoms of patients receiving long-term hemodialysis. Tracing back to the development of its relating studies, there is no accurate reason that why does people undergoing hemodialysis feel fatigued. Conclusive predictors of fatigue are still not shown up yet. Paper review indicated that the level of L-Carnitine concentration, which affect metabolism of fatty acid, had correlation with fatigue and muscle strength in this population. The serum concentration of L-Carnitine is influenced a lot by hemodialysis. When there is deficiency of energy supply, it resulted to decline of muscle strength, which increased frequency and intensity of fatigue. Hence, the purposes of this study are (1) to understand the basic condition of fatigue level, muscle and metabolism of fat and carbohydrate among hemodialysis patients, (2) to analyze correlation among muscle strength, metabolism of fat/carbohydrate, and fatigue, and (3) to understand correlations among demographic characteristics, blood test data (hemoglobin, albumin, Kt/V, urea reduction ratio(URR), blood urea nitrogen(BUN), creatinine, calcium, phosphorus, and C-reactive protein), mental and social conditions (depression, anxiety, and social support), muscle strength and fatigue, seeking further exploring predictors of muscle strength and fatigue.

The study use cross-sectional descriptive correlative design with consecutive sampling. Recruit patients from a hemodialysis unit in a medical center in north Taiwan after informed- consent. The estimated sample size is 100. To understand relationship among muscle strength, by-products of fatty acid and carbohydrate and fatigue, we collect data by measuring their muscle strength (handgrip and 30 seconds sit-to-stand), and analyzing blood test data and the structured questionnaires which included mental/social data (depression, anxiety, social support and fatigue level). Descriptive statistics, ANOVA, Pearson's correlation, Spearsman's rank correlation and stepwise regression were used to analyze the collected data. Hope this research can get advance in comprehension of cause of fatigue and improve the fatigue symptom of hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Hemodialysis Patients 2.Aged above 20 3.Consciousness: oriented

Exclusion Criteria:

* 1. Unable to complete muscle strength test or questionnaire

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients receiving regular hemodialysis thrice or twice per week
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Relationships Among Fatigue, Muscle Power and Metabolomics | 1-year study

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun Shun, PHD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan